CLINICAL TRIAL: NCT06210321
Title: Randomised Controlled Study of the Efficacy and Acceptability of a Pharmacogenetic Test in the Management of Patients Treated With Escitalopram.
Brief Title: Pharmacogenetic Testing at Community Pharmacy
Acronym: OffiGene
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chantal Csajka (Other)
Responsible Party: Sponsor-Investigator, Chantal Csajka, Professor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OffiGene01
Record Dates: First submitted 2023-03-23; First posted 2024-01-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Pharmacogenetic Testing
Keywords: Community pharmacy; Escitalopram

STUDY DESIGN:
Intervention Model Description: This study consists of two groups, an intervention group using CYP2C19 genetic information to validate escitalopram prescriptions, and a control group without using CYP2C19 genetic information.
Who Masked: Participant
Masking Description: Patients in each group will be blinded, as CYP2C19 genetic information is not given until the study is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Other): Adjustment of antidepressant treatment according to pharmacogenetic results obtained by genetic testing for cytochrome CYP 2C19 (alleles *2, *3 and *17)
  Interventions: Other: Prescription of escitalopram using pharmacogenetic testing
- Control arm (No Intervention): Delivery of escitalopram treatment as prescribed. Genetic analysis will be performed in batch at the end of the follow-up period.

INTERVENTIONS:
Other: Prescription of escitalopram using pharmacogenetic testing — Adjustment of escitalopram treatment according to pharmacogenetic results obtained by genetic testing for cytochrome CYP 2C19 (alleles *2, *3 and *17)
  Arms: Intervention arm

SUMMARY:
The purpose of this study is to assess the clinical impact of reducing treatment failure rates after using genetic information targeting CYP2C19 in validating escitalopram prescription. 5 pharmacies in the canton of Vaud (Lausanne, Switzerland) will participate in the study.

The study will also explored the ability to perform the test in community pharmacy, physician and pharmacist approval of prescription changes, patient acceptance of the test and dose changes, the economic impact of the test, the association between genetic polymorphisms and therapeutic failures and the degree of satisfaction, barriers and facilitators by stakeholders.

DETAILED DESCRIPTION:
Response to medication depends on many clinical, demographic, environmental, and genetic factors. Non-genetic factors that are often considered when prescribing treatments address not only drug-drug interactions, but also the patient's environment, comorbidities, gender, and age. Genetic factors, which are not commonly considered during prescribing except for some drugs, account for 15-30% of the variability in drug response. From a pharmacokinetic point of view, genetic polymorphisms are likely to modify drug absorption, metabolism, transport and elimination. Data from the literature indicate that the concentration profiles of many drugs are genetically influenced. It is also well known that genetic polymorphisms that alter the targeting of some drugs can alter drug response, especially in oncology.

Personalization of medicine is a fundamental approach to treating patients individually. Pilot studies to integrate pharmacogenetics into practice are already being conducted in hospitals, and some pharmacies abroad offer pharmacogenetic testing, as in Canada and Germany.

In Switzerland, a new Ordinance on Genetic Analysis Act was passed on September 23, 2022, allowing pharmacists to carry out genetic testing in the medical field.Because of the increasing evidence of the influence of CYP2C19 genetic polymorphisms on the efficacy and toxicity of escitalopram, the high prevalence of prescription of this drug in the treatment of depression, the prevalence of genetic polymorphisms in the Caucasian population (30% ultra-rapid metabolizers and 4% poor metabolizers) and the potential costs to public health, this drug was chosen as a prototype for this pilot project.

Therefore, investigators want to conduct a pilot study to evaluate the efficacy, safety, feasibility, and cost-effectiveness of pharmacy-based genetic testing as part of patient care management and identified barriers to using such tests.

ELIGIBILITY:
Inclusion Criteria:

* Must consent to participate in the study,
* Must sign consent,
* Must be able to follow and understand the study procedures,
* Initiation of escitalopram treatment for unipolar depression with or without anxiety

Exclusion Criteria:

* Other condition than depression (such as panic disorder)
* Escitalopram treatment already received
* Not able to consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-08-14 (Estimated); Study Completion 2027-08-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants in the intervention and control groups who experienced a treatment failure on escitalopram. | From enrollment to last follow-up: circa 3 months
  Number of escitalopram treatment failures in patients with escitalopram prescription based on CYP2C19 genetic testing information versus the control group prior to normal care. Treatment failure is defined here as discontinuation, dose change, or treatment change.

REFERENCES:
- [Background] Zhou Y, Ingelman-Sundberg M, Lauschke VM. Worldwide Distribution of Cytochrome P450 Alleles: A Meta-analysis of Population-scale Sequencing Projects. Clin Pharmacol Ther. 2017 Oct;102(4):688-700. doi: 10.1002/cpt.690. Epub 2017 May 26. PMID 28378927
- [Background] Eichelbaum M, Ingelman-Sundberg M, Evans WE. Pharmacogenomics and individualized drug therapy. Annu Rev Med. 2006;57:119-37. doi: 10.1146/annurev.med.56.082103.104724. PMID 16409140
- [Background] U.S. Food and Drug Administration. Table of pharmacogenomic biomarkers in drug labeling. https://www.fda.gov/drugs/science-and-research-drugs/table-pharmacogenomic-biomarkers-drug-labeling/. Accessed November, 15 2022.
- [Background] CHUV - Département oncologie. Une médecine sur mesure grâce à l'analyse génétique des tumeurs. 30.07.2018
- [Background] Veronika Litinski RD, PH. D., Boyko Kabakchiev, PH. D., Lou Carsley, Liz Garman, Gil McGowan, Gouri Mukerjee, PH. D. Pillcheck 2021 [Available from: https://www.pillcheck.ca/.
- [Background] Prof. Dr Theo Dingermann, Prof. Dr. Dieter Steinhilber. Stratipharm [cited 2022 03.06]. Available from: https://www.stratipharm.de/.
- [Background] Loi sur l'analyse génétique : renforcement de la protection contre les abus, (2022).
- [Background] Evans WE, McLeod HL. Pharmacogenomics--drug disposition, drug targets, and side effects. N Engl J Med. 2003 Feb 6;348(6):538-49. doi: 10.1056/NEJMra020526. No abstract available. PMID 12571262
- [Background] Phillips KA, Veenstra DL, Oren E, Lee JK, Sadee W. Potential role of pharmacogenomics in reducing adverse drug reactions: a systematic review. JAMA. 2001 Nov 14;286(18):2270-9. doi: 10.1001/jama.286.18.2270. PMID 11710893
- [Background] Ionova Y, Ashenhurst J, Zhan J, Nhan H, Kosinski C, Tamraz B, Chubb A. CYP2C19 Allele Frequencies in Over 2.2 Million Direct-to-Consumer Genetics Research Participants and the Potential Implication for Prescriptions in a Large Health System. Clin Transl Sci. 2020 Nov;13(6):1298-1306. doi: 10.1111/cts.12830. Epub 2020 Jul 21. PMID 32506666
- [Background] Berm EJ, Looff Md, Wilffert B, Boersma C, Annemans L, Vegter S, Boven JF, Postma MJ. Economic Evaluations of Pharmacogenetic and Pharmacogenomic Screening Tests: A Systematic Review. Second Update of the Literature. PLoS One. 2016 Jan 11;11(1):e0146262. doi: 10.1371/journal.pone.0146262. eCollection 2016. PMID 26752539